CLINICAL TRIAL: NCT06892210
Title: Comparing Hydrocortisone and Prednisolone for Acute Exacerbation of Chronic Obstructive Pulmonary Disease (AECOPD)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Copenhagen Respiratory Research (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MineraloCOP
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Methylprednisolone; Pharmaceutical Preparations; Hydrocortisone

STUDY DESIGN:
Intervention Model Description: The study is a cluster randomized controlled trial. It consists of two arms, in which patients will be randomized to receive treatment with either Hydrocortisone or Methylprednisolone.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment with Hydrocortisone. (Active Comparator): This arm will recieve a dose of 200 mg of Hydrocortisone intravenously once daily for five days.
  Interventions: Drug: Hydrocortisone
- Treatment with Methylprednisolone (Active Comparator): This arm will recieve a dose of 40 mg of Methylprednisolone intravenously once daily for five days.
  Interventions: Drug: Methylprednisolone (drug)

INTERVENTIONS:
Drug: Methylprednisolone (drug) — ATC code: H02AB06. Can be changed to Prednisolone 50 mg orally.
  Arms: Treatment with Methylprednisolone
Drug: Hydrocortisone — ATC-code: H02AB09. Can be changed to 50 mg x 4 daily orally if appropriate.
  Arms: Treatment with Hydrocortisone.

SUMMARY:
The goal of this cluster randomized controlled trial is to determine the optimal treatment for Acute Exacerbation of Chronic Obstructive Pulmonary Disease. The study compares the effects and side effects of hydrocortisone and prednisolone in patients above 40 years old diagnosed with chronic obstructive pulmonary disease with acute exacerbation. The main question is whether there is a difference in readmission for COPD excerbation or all cause mortality within thirty days.

Participants will randomized to receive treatment with either hydrocortisone or prednisolone.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥40 years
* Chronic obstructive pulmonary disease with acute exacerbation, unspecified: ICDJ44

Exclusion Criteria:

* All diagnoses that would merit treatment with a specific corticosteroid
* Pregnant or breastfeeding women
* Active tuberculosis or invasive fungal infection

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Readmission for COPD exacerbation or death from all causes | 30 days

SECONDARY OUTCOMES:
Days alive and out of hospital | 14 days
Mortality | 90 days
Readmission for COPD exacerbation | 90 days
All-cause infections | 90 days
  Defined as a new prescription of antibacterial medication.
Need for mechanical ventilation | 30 days
New onset infections | 30 days
Daily amount of insulin administered to the patient by day 7 or discharge from hospital | 7 days
Gastrointestinal bleeding | 30 days
Blood glucose levels | 7 days
  Measured at day 3 and day 7

OTHER OUTCOMES:
Procalcitonin (PCT) at baseline | 7 days
  Procalcitonin (PCT) at baseline, day 3 and day 7. If still at hospital.
C-reactive protein (CRP) at baseline | 7 days
  C-reactive protein (CRP) at baseline, day 3 and day 7. If still in hospital.
Blood eosinophil count (EOS) at baseline | 7 days
  Blood eosinophil count (EOS) at baseline, day 3 and day 7. If still in hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Ulrik Stæhr Jensen, MD, PHD, Study Director — COP:RESP

IPD SHARING:
Plan to Share IPD: Undecided
This has not yet been decided.